CLINICAL TRIAL: NCT04103177
Title: A Structured Exercise and Educational Intervention to Increase Physical Activity in Haemodialysis Patients: a Feasibility Study
Brief Title: Physical Activity in Haemodialysis Patients: a Feasibility Study
Acronym: PA-CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Helen Dawes, Director Centre for Movement, Occupational and Rehabilitation Sciences, Oxford Brookes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201762; 19/EM/0042 (Other: Research Ethics Committee- East Midlands Nottingham 1)
Record Dates: First submitted 2019-09-19; First posted 2019-09-25 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: End Stage Renal Failure on Dialysis

STUDY DESIGN:
Intervention Model Description: This pilot study will incorporate instructor led guidance of a range of chair-based exercises that focus on balance, strength, fitness, endurance and flexibility with some exercises having a cardiovascular component. These chair based exercises are drawn from programmes recommended for similar long term clinical conditions (e.g cardiovascular disease, sarcopenia, frail and elderly and renal disease) and can be performed in the clinical environment or at home.The intervention is multifaceted comprising of the following; an education booklet about PA and the chair based exercise programme, face to face instructor led support detailing the chair based exercises and instructor/nurse led motivational interviewing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): 20 participants to receive physical activity educational booklet with instructions on chair based exercises, Instructor-led training on how to perform the chair based exercises, two times a week, over a 6 week period, and motivational interviewing and prompts.
  Interventions: Other: Chair based exercises in the dialysis environment

INTERVENTIONS:
Other: Chair based exercises in the dialysis environment — Each participant will be given an educational / information booklet. It will include when the right time to engage in Physical Activity. The Chair-based Exercise Program will be the focus of the exercise intervention with written step- by-step instructions with demonstrative image of the exercises. Further details included in this booklet will include, information regarding the benefits of exercise including walking and safety measures in undertaking the exercises.
  Sports Exercise Instructor led Chair-based Exercise Programme Patients will be given Sports Exercise Instructor led training on how to perform the chair-based exercises, for 6 weeks. This will be delivered during one of the patients' dialysis sessions. The Instructor will deliver a short 10 minute session to patients and deliver safety instruction.
  Motivational interviewing Motivational interviewing will consist of discussion to encourage the participant without coercion and help them develop goals.

SUMMARY:
There is a well established link between physical inactivity and increased mortality in the general population and across many of the more common disease areas including chronic kidney disease (CKD). Patients with CKD have very high levels of morbidity and mortality and are known to have low fitness levels. Randomised controlled trials of exercise have demonstrated the benefits of physical activity for CKD patients. Despite this, physical activity levels remain low and translating these research findings into clinical practice is challenging.

This feasibility study aims to assess the feasibility and acceptability of an instructor led structured exercise programme which includes an educational component to engage and increase physical activity levels in haemodialysis patients attending the Oxford University Hospitals Trust haemodialysis unit. Consented participants will fill in a self reported physical activity questionnaire (Human Activity Profile), partake in functional mobility assessments including (Timed-Up and Go) and a chair based exercise programme. At the end of the study, participants, and nursing staff will undertake a semi-structured interview aimed at understanding acceptability of the intervention. The results of this feasibility study will then be used to inform whether a larger trial in haemodialysis patients is feasible. All questionnaires, physical activity interventions and interviews will be undertaken during routine visits to the haemodialysis unit.

DETAILED DESCRIPTION:
There is a well established link between physical inactivity and increased mortality in the general population and patients with chronic kidney disease (CKD) have low fitness levels when compared to their healthy counterparts (50% of expected norm when commencing dialysis therapy). Trials have shown that physical activity confers many physical and mental health benefits in this patient population, with improvements in fitness, walking capacity, health of the heart and quality of life; indeed, national guidelines now consider physical activity to be a cornerstone of disease management (Cochrane Collaboration 2006; Workgroup KD 2005). CKD patients have lower levels of physical activity than age-matched controls; this is particularly marked for older patients and those on dialysis. The Department of Health recommends ≥150 mins/ week of moderate intensity PA (accumulated in bouts of at least 10 minutes) for the general population (DoH UK Physical Activity Guidelines 2011). Many studies have sought to characterise the most effective forms of exercise for CKD patients. Recent attention has focussed on intradialytic cycling, with studies showing benefits not only for fitness and endurance but also muscle strength, power, and physical function. However, translating research guided physical activity programmes into routine clinical practice is challenging, requiring consideration of patients' physical and psychological barriers to exercise.

Assessing the impact of any activity programme requires comparison of health and exercise behaviours pre and post intervention. Several self-report physical activity questionnaires are available but the Human Activity Profile has been validated in CKD patients (Johansen et al. 2001). However, information obtained from patient self-reporting is subjective and prone to bias. Objective measurement devices such as accelerometers are more accurate.

Feasibility of an effective intervention to increase physical activity requires understanding of perceptions of exercise in the population of interest. In this way, the intervention can be specifically targeted to take account of perceived benefits and barriers towards physical activity and thereby increase compliance. This study will provide: 1)feasibility and acceptability of an instructor led chair based exercise programme and educational package (booklet); 2) both self-report and objective measurements of physical activity levels in a sample of haemodialysis patients. This key information will later be used to assess whether a informed large scale PA intervention study in haemodialysis patients is feasible.

ELIGIBILITY:
Inclusion Criteria:

* • Participant is willing and able to give informed consent for participation in the trial.

  * Male or Female, aged 18 years or above.
  * Undergoing regular haemodialysis (2 or 3 times per week) in the Oxford Main and Tarver Dialysis Units
  * Is able and willing to comply with all trial requirements.
  * Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Unable to give consent
* Poor dialysis compliance
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Participant with life expectancy of less than 1 month and/or receiving palliative care.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Planning to leave Oxford Dialysis units within the study trial
* Absolute contra-indications to PA including:

  * Recent significant change in resting ECG suggesting significant ischaemia, recent Myocardial Infarction within 2 days or acute cardiac event
  * Unstable angina
  * Uncontrolled cardiac arrhythmia causing symptoms or haemodynamic compromise
  * Symptomatic severe aortic stenosis
  * Uncontrolled symptomatic heart failure
  * Acute pulmonary embolus or infarction
  * Acute myocarditis or pericarditis
  * Third degree heart block
  * Suspected or know dissecting aortic aneurysm
  * Acute systemic infection, accompanied by fever, body aches or swollen lymph glands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Semi structured interviews and questionnaires targeted to determine participant acceptability of PA intervention and the people delivering it | Interviews should last no longer than an hour and will be conducted at month 3 post baseline
  Interviews with patients and staff

SECONDARY OUTCOMES:
Change is being assessed 3 metre Timed Up and Go | Change from baseline functional mobility at 6 months
  Functional activity, 1 minute to complete
Change is being assessed 10 metre walk test | Change from baseline functional mobility at 6 months
  Functional activity, 5 minutes to complete
Change is being assessed Hand grip strength | Change from baseline arm strength at 6 months
  Functional strength, 2 minutes to complete.
Change is being assessed Wrist worn accelerometery data | Change from baseline of activity at 6 months
  Accelerometers to be worn for one week at 3 time points to assess daily activity
Change is being assessed EQ-5D-3L questionnaire | Change from baseline quality of life at 6 months
  This is a self-completing short questionnaire comprising questions on the following 5 areas: mobility, self-care and daily activities. This should take no longer to complete.
Change is being assessed IPOS Renal questionnaire | Change from baseline quality of life at 6 months
  This is self-completing questionnaire comprising of 11 questions assessing renal symptoms with other items for additional concerns. 10 minutes to complete
Change is being assessed Human Activity profile questionnaire | Change from baseline of physical activity at 6 months
  This tick box questionnaire consists of 94 questions and seeks to determine the activities participants currently do. 15 minutes to complete
Falls and Fractures questionnaire | Change from baseline
  We wish to know if participants have had any falls or fractures in the last 6 months and assess baseline mobility level.
  Questions are based on Yes or No
  Referred medical falls clinic☐ Referred therapy falls clinic☐ Referred non-FLS primary care No. of falls, slips, trips in last 12 months= Indoor Gait: range from 1-2 Outdoor Gait: range from 1-2 Any Indoor falls- yes or no
  Broken bones in adult hood= Yes/No
Client Service Receipt Inventory Questionnaire | Change from baseline
  Participants will be given as short tick-box questionnaire to collect information regarding other hospitals facilities they have visited including General Practitioner visits over the last 6 months. This will exclude routine visits to haemodialysis.
  Hospital departments and services used in last 6 months- No=0 Yes=1 Use of community care services in last 6 months- No=0 Yes=1 Diagnostic tests in last 6 months- No=0 Yes=1 Use of mobility aids in last 6 months- No=0 Yes=1 Adaptations at home in last 6 months-No=0 Yes=1 Changes in informal care in last 6 months months- No=0 Yes=1 Journeys to receive care in last 6 months No=0 Yes=1 Current occupation range of 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Helen Dawes, PhD, Principal Investigator — University of Exeter
Locations (1):
- Oxford University Hospitals NHS FT, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared with other researchers in accordance with NHS Information Governance Policy (NHS Information Sharing Policy v2) and Oxford Brookes data sharing policies (Oxford Brookes IT policies). Plans for data sharing will be included in the data management plan, as well as the trial protocol. A data sharing statement will be included in the consent form and information provided in the patient information leaflet.
  Data will be pseudonymised wherever possible prior to being shared with other researchers and the information required to "decode" this data will be stored securely elsewhere, in accordance with ICH GCP guidelines. If this is not possible then consent will be obtained from participants and approval sought from the HRA prior to the trial commencing.
Supporting Information: Study Protocol
Time Frame: Time frame: Once all data analysis has taken place and the core findings have been published, they will be archived securely using Arkivum (see above). Dataset preparation will be carried out by individuals with an understanding of data management and basic statistics, with quality control provided by a further individual who is independent of the process. Researchers will be able to apply to access archived data as required.
Access Criteria: Once data has been archived in Arkivum, access will be granted to researchers in accordance with NHS and Oxford Brookes policies. Data access requests will be made via an application form detailing the specific requirements and the proposed research and publication plan, which will be reviewed against specific eligibility criteria by data custodians or by an external Independent Review Panel. Decisions about requests will be made promptly (no more than 3 months after receipt of request) and details of all data requests and their outcomes will be made publicly available (data requesters should be informed of this in advance of this).
  Funds for responsible data sharing will be requested from trial funders as part of initial trial grant applications.
URL: http://arkivum.com